CLINICAL TRIAL: NCT03479541
Title: Sensory Integration Balance Deficits in Complex mTBI: Can Early Initiation of Rehabilitation With Wearable Sensor Technology Improve Outcomes?
Brief Title: Can Early Initiation of Rehabilitation With Wearable Sensor Technology Improve Outcomes in mTBI?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Medical Research Foundation, Oregon (Other)
Responsible Party: Principal Investigator, Laurie King, Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DOD2; W81XWH-17-1-0424 (Other Grant/Funding Number: Department of Defense (DOD))
Record Dates: First submitted 2018-02-15; First posted 2018-03-27 (Actual); Results first posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Mild Traumatic Brain Injury; Balance; Distorted; Gait, Unsteady; Quality of Life; Veterans
Keywords: mild traumatic brain injury; vestibular impairment; balance and gait; dual-tasking; veterans; quality of life; rehabilitation
MeSH Terms: conditions — Brain Concussion; Gait Disorders, Neurologic | interventions — Biofeedback, Psychology

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Single-blinded design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Earlier Physical Therapy (Experimental): Within a week of enrollment and baseline testing, participants (n=80) will see a physical therapist in person twice per week for 2 weeks and once per week for 4 weeks for a total of 8 sessions over 6 weeks.
  Interventions: Behavioral: Timing of Rehabilitation
- Later Physical Therapy (Standard of Care) (Active Comparator): Participants (n=80) will wait 6 weeks after enrollment and baseline testing before starting physical therapy. Before starting physical therapy participants will be re-tested on study outcomes.
  Interventions: Behavioral: Timing of Rehabilitation
- Physical Therapy with Home Monitoring (Experimental): Participants (n=80) will start physical therapy after baseline testing and use wearable sensors during home exercise. Feedback was provided later at the next physical therapy session.
  Interventions: Behavioral: Biofeedback
- Physical Therapy (without home monitoring) (Active Comparator): Participants (n=80) will start physical therapy after baseline testing and did not use wearable sensors during home exercise. No feedback of performance was provided.
  Interventions: Behavioral: Biofeedback

INTERVENTIONS:
Behavioral: Timing of Rehabilitation — Participants in the Earlier Physical Therapy group will start physical therapy within a week of enrollment and baseline testing. Participants allocated to the Later Physical Therapy group will wait 6 weeks after enrollment and baseline testing before starting physical therapy, and re-test on study outcomes before starting physical therapy. Both groups will see a physical therapist in person twice per week for 2 weeks and once per week for 4 weeks for a total of 8 sessions over 6 weeks. Each session will last 60 minutes and consist of cardiovascular, cervical spine, and vestibular therapy exercises (static and dynamic balance). Participants will perform daily home exercises for 30 minutes with similar subcategories from the in-person sessions. Both the in-person physical therapy and home exercises will be individualized and progressive at the discretion of the physical therapist depending on the performance of the participant.
  Arms: Earlier Physical Therapy; Later Physical Therapy (Standard of Care)
Behavioral: Biofeedback — Wearable sensors measure movement during the home exercise program for later feedback.
  Arms: Physical Therapy (without home monitoring); Physical Therapy with Home Monitoring

SUMMARY:
Every year 1.7 million people sustain a traumatic brain injury (TBI) in the United States and of these, 84 % are considered mild TBI (mTBI). mTBI is common both in civilian and military populations and can be debilitating if symptoms do not resolve after injury. Balance problems are one of the most common complaints after sustaining a mTBI and often prevent individuals from returning to their previous quality of life. However, the investigators currently lack clear guidelines on when to initiate physical therapy rehabilitation and it is unclear if early physical therapy is beneficial. The investigators believe that the underlying problem of imbalance results from damage to parts of the brain responsible for interpreting sensory information for balance control. The investigators hypothesize that retraining the brain early, as opposed to months after injury, to correctly interpret sensory information will improve recovery. The investigators also believe this retraining is limited when rehabilitation exercises are performed incorrectly, and that performance feedback from wearable sensors, can improve balance rehabilitation. There are three objectives of this study: 1) to determine how the timing of rehabilitation affects outcomes after mTBI; 2) to determine if home monitoring of balance exercises using wearable sensors improves outcomes; and 3) to develop a novel feedback system using wearable sensors to provide the physical therapist information, in real-time during training, about quality of head and trunk movements during prescribed exercises. The findings from this research could be very readily adopted into military protocols for post-mTBI care and have the potential to produce better balance rehabilitation and quality of life for mTBI patients and their families.

DETAILED DESCRIPTION:
Although balance is one of the most common and debilitating complaints after mTBI, the investigators currently lack clear guidelines on when to initiate balance rehabilitation and it is unclear if early physical therapy is beneficial. There is a clear gap in clinical care guidelines after mTBI and it is unclear if initiating rehabilitation early would improve outcomes related to imbalance. Measures of imbalance are subjective and are easily overlooked as a treatable deficit. Even with rehabilitation, recovery of balance in people with mTBI is challenging, particularly in people with central vestibular and sensory integration deficits.

Although vestibular and balance rehabilitation after mTBI relies heavily on a home exercise program and repetition is essential for recovery; The slow progress in balance rehabilitation may be partially due to an inability of people with mTBI to correctly perform the prescribed rehabilitation exercises on their own. Biofeedback is a clinical technique that provides physiologic information that would otherwise be unknown to patients and may improve outcomes after mTBI. There are no commercially available systems to provide the physical therapist and/or patient objective information on the quality of head movements during training of rehabilitation tasks that involve balance and walking.

Therefore, the three objectives of this study are: 1) to determine how the timing of rehabilitation affects outcomes after mTBI; 2) to determine if home monitoring of home balance exercises using wearable sensors improves outcomes; and 3) to develop a novel feedback system using wearable sensors to provide the physical therapist information, in real-time during training, about quality of head and trunk movements during prescribed exercises.

160 individuals with subacute mTBI within 2-12 weeks of the injury will be randomly assigned to receive earlier onset of physical therapy (n=80) right away or be randomly assigned to receive later rehabilitation 6 weeks after enrollment in the standard of care physical therapy group (n=80). A subgroup of participants in the earlier physical therapy (n=40) and standard of care physical therapy (n=40) will be randomly assigned to home monitoring. The participants in the home monitoring subgroups will wear wireless sensors while completing the rehabilitation program to better inform the physical therapist of their progress.

The outcome measures will consist of a battery of self-reported questionnaires, and balance and gait measures and will be tested at Pre I (baseline), Pre 2 (6 weeks after baseline for the later physical therapy group), Post (after the intervention), and Retention (6 month follow-up). Peripheral vestibular and ocular motor assessments will occur at the baseline visit only.

The central hypothesis is that rehabilitation after mTBI is suboptimal due to late initiation of and inadequate performance of exercises that do not adequately challenge vestibular and sensory integration function. The long-term goal is to clarify best practices for the rehabilitation of balance deficits in people with mTBI by comparing earlier vs later (standard of care) initiation of physical therapy with and without wearable sensors on balance deficits after mTBI. The findings from this research could be very readily adopted into military protocols for post-mTBI care and have the potential to produce better balance rehabilitation and quality of life for mTBI patients and their families.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria will consist of being 1) 18-60 years of age; 2) having no more than minimal cognitive impairment as assessed by the Short Blessed test; 3) having a physician-diagnosed mTBI and being within 2-12 weeks of the injury; and 4) endorsing ≥1 on either balance, dizziness, nausea, headache, or vision problems on the symptom evaluation scale from the Sport Concussion Assessment Tool (SCAT 5) and a total symptom severity score ≥15.

Exclusion Criteria:

* Exclusion criteria will consist of: 1) having other musculoskeletal, neurological, or sensory deficits that could explain their dysfunction other than mTBI; 2) having moderate to severe substance use disorder within the past month; 3) experiencing severe pain during the evaluation (≥7/10 subjective rating), 4) are pregnant; and 5) are currently being treated by vestibular physical therapy; All participants will be asked to refrain from taking drugs that may influence balance including sedating antihistamines, benzodiazepines, sedatives, narcotic pain medications, and alcohol for at least 24 hours prior to testing.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 203 (Actual)
Dates: Start 2018-07-15 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Faul, M., Xu, L., Wald, M. M., & Coronado, V.G. (2010). Traumatic brain injury in the United States: Emergency Department Visits, Hospitalizations and Deaths 2002-2006. Atlanta, GA: Centers for Disease Control and Prevention, National Center for Injury Prevention and Control. https://www.cdc.gov/traumaticbraininjury/pdf/blue_book.pdf
- [Background] Pfaltz CR, Kamath R. Central compensation of vestibular dysfunction. I. Peripheral lesions. Pract Otorhinolaryngol (Basel). 1970;32(6):335-49. doi: 10.1159/000274957. No abstract available. PMID 5313795
- [Background] Shepard NT, Telian SA. Programmatic vestibular rehabilitation. Otolaryngol Head Neck Surg. 1995 Jan;112(1):173-82. doi: 10.1016/S0194-59989570317-9. PMID 7816453
- [Derived] Campbell KR, Antonellis P, Peterka RJ, Wilhelm JL, Scanlan KT, Pettigrew NC, Chen S, Parrington L, Fino PC, Chesnutt JC, Horak FB, Hullar TE, King LA. In People With Subacute Mild Traumatic Brain Injury, Earlier Physical Therapy Improved Symptoms at a Faster Rate Than Later Physical Therapy: Randomized Controlled Trial. Phys Ther. 2025 Feb 6;105(2):pzae180. doi: 10.1093/ptj/pzae180. PMID 39693261
- [Derived] Campbell KR, Scanlan KT, Wilhelm JL, Brumbach BH, Pettigrew NC, Neilson A, Parrington L, King LA. Assessment of balance in people with mild traumatic brain injury using a balance systems model approach. Gait Posture. 2023 Feb;100:107-113. doi: 10.1016/j.gaitpost.2022.12.005. Epub 2022 Dec 7. PMID 36516644
- [Derived] Campbell KR, Wilhelm JL, Pettigrew NC, Scanlan KT, Chesnutt JC, King LA. Implementation and Adoption of Telerehabilitation for Treating Mild Traumatic Brain Injury. J Neurol Phys Ther. 2022 Oct 1;46(4):E1-E10. doi: 10.1097/NPT.0000000000000409. Epub 2022 Jun 6. PMID 35666882
- [Derived] Parrington L, Jehu DA, Fino PC, Stuart S, Wilhelm J, Pettigrew N, Murchison CF, El-Gohary M, VanDerwalker J, Pearson S, Hullar T, Chesnutt JC, Peterka RJ, Horak FB, King LA. The Sensor Technology and Rehabilitative Timing (START) Protocol: A Randomized Controlled Trial for the Rehabilitation of Mild Traumatic Brain Injury. Phys Ther. 2020 Apr 17;100(4):687-697. doi: 10.1093/ptj/pzaa007. PMID 31951263

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were screened for eligibility (n=2522) and recruited from institutional and local clinics in the Portland Metropolitan area. Recruitment and enrollment started in July 2018 and ended in March of 2023.
Pre-assignment Details: In-person physical therapy (PT) stopped March 2020 due to COVID-19. From April 2020 to September 2020, 18 participants were enrolled in the study and received telerehabilitation. However, these participants were not included in further analyses due to differences from the in-person PT sessions. Although there are 4 arms to the study, those included in the early and late PT groups were the same people in the home monitoring groups. Therefore, the total included is 203 (not 406).
Groups:
- Earlier Physical Therapy: Within a week of enrollment and baseline testing, participants will see a physical therapist in person twice per week for 2 weeks and once per week for 4 weeks for a total of 8 sessions over 6 weeks. Each physical therapy session will last 60 minutes and consist of cardiovascular exercise, cervical spine exercises, and vestibular therapy exercises (static and dynamic balance). Participants will perform daily home exercises for approximately 30 minutes with similar subcategories from the in-person physical therapy sessions. Both the in-person physical therapy and home exercises will be individualized and progressive in the sense that each exercise can increase the level of difficulty at the discretion of the physical therapist depending on the performance of the participant.
- Later Physical Therapy (Standard of Care): Participants will wait 6 weeks after enrollment and baseline testing before starting physical therapy. Before starting physical therapy participants will be re-tested on study outcomes. After waiting, participants will see a physical therapist in person twice per week for 2 weeks and once per week for 4 weeks for a total of 8 sessions over 6 weeks. Each physical therapy session will last 60 minutes and consist of cardiovascular exercise, cervical spine exercises, and vestibular therapy exercises (static and dynamic balance). Participants perform daily home exercises for approximately 30 minutes with similar subcategories from the in-person physical therapy sessions. Both the in-person physical therapy and home exercises will be individualized and progressive in the sense that each exercise can increase the level of difficulty at the discretion of the physical therapist depending on the performance of the participant.
- Physical Therapy With Home Monitoring: Wearable sensors were worn during home exercises and biofeedback was reviewed in the next physical therapy appointment.
- Physical Therapy (Without Home Monitoring): Home exercise was completed without wearable sensors, and biofeedback was not given on home exercise performance.
Period: Early and Late Physical Therapy
Arm/Group | Earlier Physical Therapy | Later Physical Therapy (Standard of Care) | Physical Therapy With Home Monitoring | Physical Therapy (Without Home Monitoring)
Started (Number of Participants Randomized) | 82 | 121 | 0 | 0
Started Physical Therapy | 75 | 81 | 0 | 0
Completed Post-Physical Therapy Assessments | 63 | 63 | 0 | 0
Completed | 63 | 63 | 0 | 0
Not Completed | 19 | 58 | 0 | 0
Not completed — Lost to Follow-up | 2 | 18 | 0 | 0
Not completed — Withdrawal by Subject | 15 | 32 | 0 | 0
Not completed — Early Termination - PI Decision | 2 | 8 | 0 | 0
Period: Home Monitoring
Arm/Group | Earlier Physical Therapy | Later Physical Therapy (Standard of Care) | Physical Therapy With Home Monitoring | Physical Therapy (Without Home Monitoring)
Started | 0 | 0 | 93 | 110
Started Physical Therapy | 0 | 0 | 73 | 83
Completed Post-Physical Therapy Assessments | 0 | 0 | 64 | 62
Completed | 0 | 0 | 64 | 62
Not Completed | 0 | 0 | 29 | 48
Not completed — Lost to Follow-up | 0 | 0 | 8 | 12
Not completed — Withdrawal by Subject | 0 | 0 | 17 | 30
Not completed — Early Termination - PI Decision | 0 | 0 | 4 | 6

BASELINE CHARACTERISTICS:
Population: One participant counted twice from the earlier physical therapy group in participant flow. They enrolled then were terminated due to re-injury then were later re-enrolled into the study with a new ID. The terminated and then re-enrolled participant's baseline demographics are presented based on the most recent injury.
Groups:
- Total: Total of all reporting groups
Arm/Group | Earlier Physical Therapy | Later Physical Therapy (Standard of Care) | Total
Number analyzed (Participants) | 81 | 121 | 202
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.6 (11.6) | 36.0 (11.2) | 35.9 (11.3)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex/Gender: Male | 18 | 20 | 38
  Sex/Gender: Female | 63 | 96 | 159
  Sex/Gender: Other | 0 | 5 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 4
  Black or African American | 1 | 1 | 2
  White | 65 | 98 | 163
  More than one race | 5 | 13 | 18
  Unknown or Not Reported | 5 | 3 | 8
Region of Enrollment [Number; unit: participants]
  United States | 81 | 121 | 202
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 25.1 (4.9) | 27.3 (8.0) | 26.4 (7.0)
Days Since Injury at Enrollment [Mean (Standard Deviation); unit: days] | 45.9 (20.1) | 45.4 (22.4) | 45.6 (21.5)
Injury Mechanism [Count of Participants; unit: Participants]
  bike-related | 3 | 6 | 9
  fall | 17 | 23 | 40
  motor vehicle accident | 24 | 47 | 71
  other | 19 | 28 | 47
  sport-related | 18 | 17 | 35
mild traumatic brain injury (mTBI) History [Count of Participants; unit: Participants]
  No | 43 | 57 | 100
  Yes | 38 | 64 | 102

OUTCOME MEASURES:

1. Primary Outcome: Dizziness Handicap Inventory (DHI)
Description: Self-rated questionnaire for dizziness impairment rated on a 3-point scale (0: no; 2: sometimes; 4: always) with a maximum score of 100. Higher scores indicate worse outcome.
Time Frame: Earlier Physical Therapy (PT) Group: Pre (week 0) and Post Physical Therapy (week 7) / Later PT Group: Baseline (week 0), Pre (week 7), and Post Physical Therapy (week 14)
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Earlier Physical Therapy: Within a week of enrollment and baseline testing, participants will see a physical therapist in person twice per week for 2 weeks and once per week for 4 weeks for a total of 8 sessions over 6 weeks. Each physical therapy session will last 60 minutes and consist of cardiovascular exercise, cervical spine exercises, and vestibular therapy exercises (static and dynamic balance). Participants will perform daily home exercises for approximately 30 minutes with similar subcategories from the in-person physical therapy sessions. Both the in-person physical therapy and home exercises will be individualized and progressive in the sense that each exercise can increase the level of difficulty at the discretion of the physical therapist depending on the performance of the participant.
  Two sub-arms include "Vestibular Rehabilitation" n=40, and "Vestibular Rehabilitation with Home Monitoring" n=40
  The group allocated to vestibular rehabilitation with home monitoring will perform the vestibular home exercises while wearing one wireless sensor on the head and one on the sternum. When the participant brings the sensors into the physical therapy session each week, the physical therapist will examine the sensor data and likely make a more informed decision as to whether or not to increase the level of difficulty of the exercises.
- Later Physical Therapy (Standard of Care): Participants will wait 6 weeks after enrollment and baseline testing before starting physical therapy. Before starting physical therapy participants will be re-tested on study outcomes. After waiting, participants will see a physical therapist in person twice per week for 2 weeks and once per week for 4 weeks for a total of 8 sessions over 6 weeks. Each physical therapy session will last 60 minutes and consist of cardiovascular exercise, cervical spine exercises, and vestibular therapy exercises (static and dynamic balance). Participants perform daily home exercises for approximately 30 minutes with similar subcategories from the in-person physical therapy sessions. Both the in-person physical therapy and home exercises will be individualized and progressive in the sense that each exercise can increase the level of difficulty at the discretion of the physical therapist depending on the performance of the participant.
  Two sub-arms include "Vestibular Rehabilitation" n=40, and "Vestibular Rehabilitation with Home Monitoring" n=40
  The group allocated to vestibular rehabilitation with home monitoring will perform the vestibular home exercises while wearing one wireless sensor on the head and one on the sternum. When the participant brings the sensors into the physical therapy session each week, the physical therapist will examine the home data and likely make a more informed decision as to whether or not to increase the level of difficulty of the exercises.
- Physical Therapy With Home Monitoring: Participants started physical therapy after baseline testing and used wearable sensors during home exercises. Feedback was provided later at the next physical therapy session.
- Physical Therapy (Without Home Monitoring): Participants started physical therapy after baseline testing and did not use wearable sensors during home exercises. No feedback of performance was provided.
Arm/Group | Earlier Physical Therapy | Later Physical Therapy (Standard of Care) | Physical Therapy With Home Monitoring | Physical Therapy (Without Home Monitoring)
Number analyzed (Participants) | 82 | 121 | 93 | 110
score on a scale
  Estimated Mean at Enrollment | 29.2 [25.4 to 33.0] | 34.9 [31.4 to 38.4] | 33.3 [29.5 to 37.1] | 32.1 [28.3 to 35.9]
  Estimated Change per Day | -0.202 [-0.272 to -0.132] | -0.105 [-0.137 to -0.073] | -0.133 [-0.177 to -0.090] | -0.102 [-0.145 to -0.060]
Statistical Analysis 1: Comparison: Earlier Physical Therapy vs Later Physical Therapy (Standard of Care); Test type: Other — Linear mixed effect model containing fixed effects for group (earlier or later), time since injury, and group x time since injury interaction with random intercepts, covariates (age, gender, and Initial SCAT symptom severity total score), and inverse probability weights. Later Physical Therapy Group served as the reference; p = 0.013, Mixed Models Analysis — a priori threshold p < 0.05; Slope = -0.097, 95% CI 2-sided [-0.173 to -0.020] — The slope estimate is the group difference (Early Physical Therapy Group - Later Physical Therapy Group) in change per day per day (the interaction effect of the mixed model analysis)

2. Secondary Outcome: Neurobehavioral Symptom Inventory (NSI)
Description: Self-rated questionnaire (~5 minutes) for symptom severity on a scale from 0 (none) to 4 (very severe) with a maximum score of 88. High scores indicate worse outcomes.
Time Frame: Earlier PT Group: Pre (week 0) and Post Physical Therapy (week 7) / Later PT Group: Baseline (week 0), Pre (week 7), and Post Physical Therapy (week 14)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Earlier Physical Therapy | Later Physical Therapy (Standard of Care) | Physical Therapy With Home Monitoring | Physical Therapy (Without Home Monitoring)
Number analyzed (Participants) | 82 | 121 | 93 | 110
score on a scale
  Estimated Mean at Enrollment | 39.1 [36.3 to 41.9] | 43.5 [41.1 to 45.9] | 42.7 [39.9 to 45.5] | 40.9 [38.3 to 43.5]
  Estimated Change per Day | -0.259 [-0.311 to -0.207] | -0.186 [-0.210 to -0.162] | -0.23 [-0.235 to -0.170] | -0.189 [-0.221 to -0.158]
Statistical Analysis 1: Comparison: Earlier Physical Therapy vs Later Physical Therapy (Standard of Care); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.013, Mixed Models Analysis — a priori threshold p < 0.05; Slope = -0.073, 95% CI 2-sided [-0.130 to -0.016] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Quality of Life After Brain Injury (QOLIBRI)
Description: Self-rated questionnaire for quality of life questioning satisfaction on a scale from 0 (not at all) to 4 (very). Scores are transformed to a scale of 0 to 100. Lower scores indicate worse outcomes.
Time Frame: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Percent
Arm/Group | Earlier Physical Therapy | Later Physical Therapy (Standard of Care) | Physical Therapy With Home Monitoring | Physical Therapy (Without Home Monitoring)
Number analyzed (Participants) | 82 | 121 | 93 | 110
Percent
  Estimated Mean at Enrollment | 49.7 [46.5 to 52.9] | 45.7 [43.1 to 48.3] | 47.9 [44.6 to 51.2] | 46.8 [44.2 to 49.4]
  Estimated Change per Day | 0.277 [0.209 to 0.345] | 0.179 [0.148 to 0.210] | 0.201 [0.159 to 0.242] | 0.192 [0.152 to 0.232]
Statistical Analysis 1: Comparison: Earlier Physical Therapy vs Later Physical Therapy (Standard of Care); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.010, Mixed Models Analysis — a priori threshold p < 0.05; Slope = 0.098, 95% CI 2-sided [0.024 to 0.173] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Patient Global Impression of Change (PGIC)
Description: This single questionnaire will ask the participant to rate how they perceive their health has changed over the course of treatment. Scores range from 1 to 7 with lower scores indicating worse performance.
Time Frame: Earlier PT Group: Post PT (week 7) / Later PT Group: Post PT (week 14)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Earlier Physical Therapy | Later Physical Therapy (Standard of Care) | Physical Therapy With Home Monitoring | Physical Therapy (Without Home Monitoring)
Number analyzed (Participants) | 63 | 63 | 64 | 62
score on a scale | 6 [5 to 7] | 6 [5 to 7] | 6 [5 to 7] | 6 [5 to 7]
Statistical Analysis 1: Comparison: Earlier Physical Therapy vs Later Physical Therapy (Standard of Care); Test type: Other; p = 0.5158, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Return to Activity Question
Description: One question asking participants how recovered they feel on a 0 (not at all recovered) to 100% (fully recovered and returned to pre-injury level) scale. Lower scores indicate worse outcomes.
Time Frame: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Percent (%)
Arm/Group | Earlier Physical Therapy | Later Physical Therapy (Standard of Care) | Physical Therapy With Home Monitoring | Physical Therapy (Without Home Monitoring)
Number analyzed (Participants) | 82 | 121 | 93 | 110
Percent (%)
  Estimated Mean at Enrollment | 59.8 [55.9 to 63.7] | 54.2 [50.4 to 58.1] | 54.1 [48.9 to 58.9] | 58.5 [54.8 to 62.2]
  Estimated Change per Day | 0.277 [0.182 to 0.372] | 0.236 [0.192 to 0.281] | 0.266 [0.208 to 0.324] | 0.224 [0.169 to 0.279]
Statistical Analysis 1: Comparison: Earlier Physical Therapy vs Later Physical Therapy (Standard of Care); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.450, Mixed Models Analysis — a priori threshold p < 0.05; Slope = 0.0404, 95% CI 2-sided [-0.0648 to 0.146] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Dynamic Visual Acuity (DVA)
Description: Physical assessment that assesses gaze stability during head rotations (horizontal and vertical) relative to head-stationary visual acuity. Higher scores indicate worse outcome.
Time Frame: Earlier PT Group: Pre (week 0) and Post Physical Therapy (week 7) / Later PT Group: Pre (week 7), and Post Physical Therapy (week 14)
Measure: Least Squares Mean (95% Confidence Interval); unit: lines lost from static visual acuity
Arm/Group | Earlier Physical Therapy | Later Physical Therapy (Standard of Care) | Physical Therapy With Home Monitoring | Physical Therapy (Without Home Monitoring)
Number analyzed (Participants) | 74 | 79 | 72 | 80
lines lost from static visual acuity
  Pre Physical Therapy Horizonal DVA Lines Lost | 1.1 [0.5 to 1.6] | 1.3 [0.7 to 1.8] | 1.4 [1.0 to 1.8] | 1.4 [1.1 to 1.7]
  Post Physical Therapy Horizonal DVA Lines Lost | 0.8 [0.2 to 1.4] | 0.8 [0.3 to 1.3] | 0.9 [0.7 to 1.2] | 1.1 [0.8 to 1.5]
  Pre Physical Therapy Vertical DVA Lines Lost | 1.3 [0.8 to 1.8] | 1.1 [0.7 to 1.6] | 1.5 [1.0 to 1.9] | 1.2 [1.0 to 1.4]
  Post Physical Therapy Vertical DVA Lines Lost | 0.6 [0.1 to 1.2] | 0.9 [0.4 to 1.4] | 0.9 [0.7 to 1.2] | 0.9 [0.6 to 1.2]
Statistical Analysis 1: Comparison: Earlier Physical Therapy vs Later Physical Therapy (Standard of Care); Analysis for Horizontal DVA Lines Lost; Test type: Other — Linear mixed effect model containing fixed effects for group (earlier or later), time point (pre-physical therapy and post-physical therapy), and group x time point injury interaction with random intercepts, covariates (age, gender, Initial SCAT symptom severity total score, and days since injury before physical therapy), and inverse probability weights. Later Physical Therapy Group and pre-physical therapy time point served as the reference. Values were log-transformed for model assumptions; p = 0.6039, Mixed Models Analysis — a priori threshold p < 0.05; Slope = 0.05353, 95% CI 2-sided [-0.1503 to 0.2574] — The slope estimate is the group difference (Early Physical Therapy Group - Later Physical Therapy Group) in change from pre-physical therapy to post-physical therapy time points (the interaction effect of the mixed model analysis)
Statistical Analysis 2: Comparison: Earlier Physical Therapy vs Later Physical Therapy (Standard of Care); Analysis for Vertical DVA Lines Lost; Test type: Other — Linear mixed effect model containing fixed effects for group (earlier or later), time point (pre-physical therapy and post-physical therapy), and group x time point injury interaction with random intercepts, covariates (age, gender, Initial SCAT symptom severity total score, and days since injury before physical therapy), and inverse probability weights. Later Physical Therapy Group and pre-physical therapy time point served as the references. Values were log-transformed for model assumptions; p = 0.0414, Mixed Models Analysis — a priori threshold p < 0.05; Slope = -0.235, 95% CI 2-sided [-0.461 to -0.0093] — [estimate comment as in outcome 6, analysis 1]

7. Secondary Outcome: Vestibular/Ocular-Motor Screening (VOMS) Tool
Description: Physical assessment (~10 minutes) to assess the function of the vestibular- and ocular-motor system, and clinically reporting symptoms of headache, dizziness, nausea, and fogginess during each visual task on a 10-point scale (0: no symptoms; 10 severe symptoms). The total symptom provocation change scores range from 0 to 280. High scores indicate worse outcomes.
Time Frame: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Earlier Physical Therapy | Later Physical Therapy (Standard of Care) | Physical Therapy With Home Monitoring | Physical Therapy (Without Home Monitoring)
Number analyzed (Participants) | 82 | 121 | 93 | 110
score on a scale
  Estimated Mean at Enrollment | 14.4 [11.7 to 17.1] | 14.6 [12.6 to 16.6] | 14.9 [12.5 to 17.2] | 14.3 [11.8 to 16.8]
  Estimated Change per Day | -0.131 [-0.188 to -0.074] | -0.103 [-0.129 to -0.077] | -0.091 [-0.125 to -0.056] | -0.116 [-0.149 to -0.083]
Statistical Analysis 1: Comparison: Earlier Physical Therapy vs Later Physical Therapy (Standard of Care); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.387, Mixed Models Analysis — a priori threshold p < 0.05; Slope = -0.028, 95% CI 2-sided [-0.090 to 0.035] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Mini-Balance Evaluation Systems Test (Mini-BESTest)
Description: Physical assessment (~20 minutes) to quantify balance and clinically scored on a 3-point scale (0: severe; 2: normal) with a maximum score of 28. Lower scores indicate worse outcomes.
Time Frame: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Earlier Physical Therapy | Later Physical Therapy (Standard of Care) | Physical Therapy With Home Monitoring | Physical Therapy (Without Home Monitoring)
Number analyzed (Participants) | 82 | 121 | 93 | 110
score on a scale
  Estimated Mean at Enrollment | 24.8 [24.3 to 25.3] | 24.4 [24.0 to 24.8] | 24.4 [23.8 to 24.9] | 24.7 [24.3 to 25.1]
  Estimated Change per Day | 0.019 [0.009 to 0.029] | 0.011 [0.006 to 0.015] | 0.011 [0.005 to 0.017] | 0.013 [0.008 to 0.019]
Statistical Analysis 1: Comparison: Earlier Physical Therapy vs Later Physical Therapy (Standard of Care); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.135, Mixed Models Analysis — a priori threshold p < 0.05; Slope = 0.008, 95% CI 2-sided [-0.003 to 0.019] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Modified Balance Error Scoring System (mBESS)
Description: Physical assessment (~5 min) that is clinically scored on a scale from 0-10 (0: no errors; 10: 10 or more errors) for each of the three conditions. High scores indicate worse outcomes.
Time Frame: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Earlier Physical Therapy | Later Physical Therapy (Standard of Care) | Physical Therapy With Home Monitoring | Physical Therapy (Without Home Monitoring)
Number analyzed (Participants) | 82 | 121 | 93 | 110
score on a scale
  Estimated Mean at Enrollment | 6.1 [4.9 to 7.4] | 6.6 [5.5 to 7.6] | 6.6 [5.2 to 7.9] | 6.2 [5.2 to 7.3]
  Estimated Change per Day | -0.0229 [-0.0459 to 0.00021] | -0.0122 [-0.0226 to -0.0018] | 0.0003 [-0.0130 to 0.0135] | -0.024 [-0.037 to -0.011]
Statistical Analysis 1: Comparison: Earlier Physical Therapy vs Later Physical Therapy (Standard of Care); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.406, Mixed Models Analysis — a priori threshold p < 0.05; Slope = -0.0107, 95% CI 2-sided [-0.0360 to 0.0146]; The slope estimate is the group difference (Early Physical Therapy Group - Later Physical Therapy Group) in change per day per day (the interaction effect of the mixed model analysis)

10. Secondary Outcome: Automated Neuropsychological Assessment Metrics (ANAM)
Description: 20-minute Computer-based test of cognition. Composite scores range from -4 to +4. Lower scores indicate worse outcome.
Time Frame: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Earlier Physical Therapy | Later Physical Therapy (Standard of Care) | Physical Therapy With Home Monitoring | Physical Therapy (Without Home Monitoring)
Number analyzed (Participants) | 82 | 121 | 93 | 110
score on a scale
  Estimated Mean at Enrollment | -0.730 [-0.933 to -0.527] | -0.732 [-0.922 to -0.543] | -0.787 [-0.985 to -0.588] | -0.685 [-0.892 to -0.478]
  Estimated Change per Day | 0.00647 [0.00243 to 0.0105] | 0.00256 [0.000716 to 0.00440] | 0.0028 [0.0003 to 0.0053] | 0.0034 [0.0011 to 0.0057]
Statistical Analysis 1: Comparison: Earlier Physical Therapy vs Later Physical Therapy (Standard of Care); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.083, Mixed Models Analysis — a priori threshold p < 0.05; Slope = 0.00391, 95% CI 2-sided [-0.00052 to 0.00835] — [estimate comment as in outcome 1, analysis 1]

11. Secondary Outcome: Instrumented Sway
Description: Participants stand with feet together with eyes closed on a firm (EcFi) and Foam (EcFo) surface for 30 seconds. An inertial sensor around the waist measures the sway area. Larger areas indicate worse performance.We generated inverse probability weights using data from all subjects, thus the overall number of participants (not the number of participants without missing values) as the overall participants analyzed.
Time Frame: as for outcome 2
Population: Two participants fell during EcFo test making the sway area invalid.
Measure: Mean (95% Confidence Interval); unit: m^4/s^2
Arm/Group | Earlier Physical Therapy | Later Physical Therapy (Standard of Care) | Physical Therapy With Home Monitoring | Physical Therapy (Without Home Monitoring)
Number analyzed (Participants) | 82 | 121 | 93 | 110
m^4/s^2
  Estimated Mean EcFi Sway Area at Enrollment | 0.160 [0.128 to 0.192] | 0.237 [0.160 to 0.314] | 0.215 [0.145 to 0.286] | 0.198 [0.129 to 0.267]
  Estimated EcFi Sway Area Change per Day | -0.006 [-0.010 to -0.001] | -0.003 [-0.005 to -0.001] | -0.0004 [-0.0013 to 0.0005] | -0.0008 [-0.0017 to 0.0001]
  Estimated Mean EcFo Sway Area at Enrollment | 0.816 [0.394 to 1.238] | 0.654 [0.546 to 0.762] | 0.687 [0.554 to 0.820] | 0.747 [0.419 to 1.075]
  Estimated EcFo Sway Area | -0.008 [-0.011 to -0.005] | -0.003 [-0.004 to -0.001] | -0.0021 [-0.0041 to -0.0002] | -0.0032 [-0.0051 to -0.0013]
Statistical Analysis 1: Comparison: Earlier Physical Therapy vs Later Physical Therapy (Standard of Care); Analysis for EcFi condition; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.240, Mixed Models Analysis — a priori threshold p < 0.05; Slope = -0.003, 95% CI 2-sided [-0.007 to 0.002] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Earlier Physical Therapy vs Later Physical Therapy (Standard of Care); Analysis for EcFo condition; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.003, Mixed Models Analysis — a priori threshold p < 0.05; Slope = -0.005, 95% CI 2-sided [-0.009 to -0.002] — [estimate comment as in outcome 1, analysis 1]

12. Secondary Outcome: Complex Navigation Task
Description: Physical assessment using wearable inertial sensors to quantify the average time to navigate a lap of a complex course (total 8 laps). Participants walk at a self-selected pace around the course under single-task and dual-task auditory Stroop conditions. Longer lap times indicate worse outcomes.
Time Frame: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Seconds
Arm/Group | Earlier Physical Therapy | Later Physical Therapy (Standard of Care) | Physical Therapy With Home Monitoring | Physical Therapy (Without Home Monitoring)
Number analyzed (Participants) | 82 | 121 | 93 | 110
Seconds
  Estimated Mean Single Task Average Lap Time at Enrollment | 14.78 [14.16 to 15.39] | 15.30 [14.85 to 15.75] | 14.94 [14.36 to 15.52] | 15.22 [14.72 to 15.73]
  Estimated Single Task Average Lap Time Change per Day | -0.0322 [-0.0421 to -0.0223] | -0.0210 [-0.0253 to -0.0168] | -0.022 [-0.028 to -0.0165] | -0.024 [-0.030 to -0.019]
  Estimated Mean Auditory Stroop Task Average Lap Time at Enrollment | 14.76 [14.19 to 15.34] | 15.40 [14.92 to 15.88] | 14.99 [14.38 to 15.60] | 15.27 [14.77 to 15.78]
  Estimated Auditory Stroop Task Average Lap Time Change per Day | -0.0300 [-0.0393 to -0.0208] | -0.0190 [-0.0230 to -0.0150] | -0.022 [-0.027 to -0.017] | -0.022 [-0.027 to -0.016]
Statistical Analysis 1: Comparison: Earlier Physical Therapy vs Later Physical Therapy (Standard of Care); Analysis for Single Task Average Lap Time; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.042, Mixed Models Analysis — a priori threshold p < 0.05; Slope = -0.0112, 95% CI 2-sided [-0.0219 to -0.0004] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Earlier Physical Therapy vs Later Physical Therapy (Standard of Care); Analysis for Auditory Stroop Average Lap Time; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0311, Mixed Models Analysis — a priori threshold p < 0.05; Slope = -0.0111, 95% CI 2-sided [-0.0211 to -0.0010] — [estimate comment as in outcome 1, analysis 1]

13. Secondary Outcome: Instrumented Walking: Gait Speed
Description: Physical assessment using wearable inertial sensors to quantify gait kinematics when walking at a self-selected pace in a straight line (9m) with and without the auditory Stroop. Gait speed at enrollment (m/s). Slower gait speeds and slower turning velocity indicate worse outcomes.
Time Frame: as for outcome 2
Population: 1 Participant from the Later PT group was excluded from Single Task 180 Deg Turn Velocity because of not following directions correctly.
Measure: Mean (95% Confidence Interval); unit: m/s
Arm/Group | Earlier Physical Therapy | Later Physical Therapy (Standard of Care) | Physical Therapy With Home Monitoring | Physical Therapy (Without Home Monitoring)
Number analyzed (Participants) | 82 | 121 | 93 | 110
m/s
  Estimated Mean Single Task Gait Speed at Enrollment | 1.313 [1.279 to 1.348] | 1.255 [1.225 to 1.286] | 1.289 [1.252 to 1.326] | 1.283 [1.251 to 1.341]
  Estimated Change in Single Task Gait Speed per Day | 0.00083 [0.00030 to 0.00136] | 0.00054 [0.00031 to 0.00077] | 0.00062 [0.00030 to 0.00093] | 0.00063 [0.00032 to 0.00093]
  Estimated Mean Auditory Stroop Gait Speed at Enrollment | 1.277 [1.243 to 1.311] | 1.227 [1.195 to 1.259] | 1.244 [1.204 to 1.284] | 1.263 [1.231 to 1.295]
  Estimated Change in Auditory Stroop Gait Speed per Day | 0.00083 [0.00032 to 0.00134] | 0.00049 [0.00026 to 0.00071] | 0.00058 [0.00028 to 0.00089] | 0.00060 [0.00030 to 0.00089]
Statistical Analysis 1: Comparison: Earlier Physical Therapy vs Later Physical Therapy (Standard of Care); Analysis for Single Task Gait Speed; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.3226, Mixed Models Analysis — a priori threshold p < 0.05; Slope = 0.00029, 95% CI 2-sided [-0.0003 to 0.00087] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Earlier Physical Therapy vs Later Physical Therapy (Standard of Care); Analysis for Auditory Stroop Gait Speed; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.2218, Mixed Models Analysis — a priori threshold p < 0.05; Slope = 0.00035, 95% CI 2-sided [-0.0002 to 0.00090]; [other analysis details as in outcome 9, analysis 1]

14. Secondary Outcome: Instrumented Walking: 180 Degree Turn Velocity
Description: Physical assessment using wearable inertial sensors to quantify gait kinematics when walking at a self-selected pace in a straight line (9m) with and without the auditory Stroop. Measure: 180-degree turning speed. Slower turning velocities indicate worse outcomes. We generated inverse probability weights using data from all subjects, thus the overall number of participants (not the number of participants without missing values) as the overall participants analyzed.
Time Frame: as for outcome 2
Population: as for outcome 13
Measure: Mean (95% Confidence Interval); unit: degrees per second
Arm/Group | Earlier Physical Therapy | Later Physical Therapy (Standard of Care) | Physical Therapy With Home Monitoring | Physical Therapy (Without Home Monitoring)
Number analyzed (Participants) | 82 | 121 | 93 | 110
degrees per second
  Estimated Mean Single Task 180 Degree Turn Velocity at Enrollment | 208.22 [199.42 to 217.03] | 194.78 [187.72 to 201.84] | 201.2 [191.6 to 210.7] | 199.4 [192.3 to 206.5]
  Estimated Change in Single Task 180 Degree Turn Velocity per Day | 0.261 [0.0999 to 0.422] | 0.100 [0.0275 to 0.173] | 0.1263 [0.0153 to 0.2372] | 0.1841 [0.0770 to 0.2911]
  Estimated Mean Auditory Stroop 180 Degree Turn Velocity at Enrollment | 204.23 [195.82 to 212.64] | 193.13 [185.54 to 200.73] | 197.0 [187.6 to 206.3] | 198.2 [190.7 to 205.8]
  Estimated Change in Auditory Stroop 180 Degree Turn Velocity per Day | 0.306 [0.152 to 0.461] | 0.0897 [0.0211 to 0.158] | 0.1801 [0.0904 to 0.2697] | 0.1099 [0.0231 to 0.1967]
Statistical Analysis 1: Comparison: Earlier Physical Therapy vs Later Physical Therapy (Standard of Care); Analysis for Single Task 180 Degree Turn Velocity; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0742, Mixed Models Analysis — a priori threshold p < 0.05; Slope = 0.161, 95% CI 2-sided [-0.0159 to 0.338] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Earlier Physical Therapy vs Later Physical Therapy (Standard of Care); Analysis for Auditory Stroop 180 Degree Turn Velocity; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0121, Mixed Models Analysis — a priori threshold p < 0.05; Slope = 0.217, 95% CI 2-sided [0.0480 to 0.385] — [estimate comment as in outcome 1, analysis 1]

15. Secondary Outcome: Instrumented Walking: Percentage of Double Support of Gait Cycle
Description: Physical assessment using wearable inertial sensors to quantify gait kinematics when walking at a self-selected pace in a straight line (9m) with and without the auditory Stroop. Percentage of gait cycle in double support were the outcome measure. Larger percentages of double support time indicate worse outcomes.
Time Frame: as for outcome 2
Population: as for outcome 13
Measure: Mean (95% Confidence Interval); unit: % of Gait Cycle
Arm/Group | Earlier Physical Therapy | Later Physical Therapy (Standard of Care) | Physical Therapy With Home Monitoring | Physical Therapy (Without Home Monitoring)
Number analyzed (Participants) | 82 | 121 | 93 | 110
% of Gait Cycle
  Estimated Mean Single Task Percentage of Double Support of Gait Cycle at Enrollment | 19.18 [18.57 to 19.79] | 20.08 [19.44 to 20.72] | 19.88 [19.16 to 20.59] | 19.59 [18.94 to 20.23]
  Estimated Change in Single Task Percentage of Double Support of Gait Cycle per Day | -0.0021 [-0.0104 to 0.00614] | -0.0027 [-0.0063 to 0.00082] | -0.0041 [-0.0089 to 0.00068] | -0.0015 [-0.0061 to 0.0032]
  Estimated Mean Auditory Stroop Percentage of Double Support of Gait Cycle at Enrollment | 19.77 [19.14 to 20.39] | 20.59 [19.92 to 21.26] | 20.61 [19.85 to 21.36] | 19.96 [19.31 to 20.61]
  Estimated Change in Auditory Stroop Percentage of Double Support of Gait Cycle per Day | -0.00278 [-0.0117 to 0.00612] | -0.0018 [-0.0057 to 0.00205] | -0.0029 [-0.0079 to 0.0020] | -0.0022 [-0.0071 to 0.0026]
Statistical Analysis 1: Comparison: Earlier Physical Therapy vs Later Physical Therapy (Standard of Care); Analysis for Single Task Percentage of Double Support Time of Gait Cycle; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.8906, Mixed Models Analysis — a priori threshold p < 0.05; Slope = 0.00063, 95% CI 2-sided [-0.0084 to 0.00961] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Earlier Physical Therapy vs Later Physical Therapy (Standard of Care); Analysis for Auditory Stroop Percentage of Double Support Time of Gait Cycle; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.8447, Mixed Models Analysis — a priori threshold p < 0.05; Slope = -0.0010, 95% CI 2-sided [-0.0107 to 0.00874] — [estimate comment as in outcome 1, analysis 1]

16. Secondary Outcome: Central Sensorimotor Integration (CSMI) Test: Visual and Vestibular Weighting
Description: Physical assessment (~45 min) to quantify sway response from a pseudo-random rotating visual surround stimulus on a fixed surface with eyes open (VS/EO) or from combined rotating visual surround and stance surface stimuli (SS+VS/EO) to calculate sensory weighting. This outcome is unitless for the weights as they are percentage values (0-1). We generated inverse probability weights using data from all subjects, thus the overall number of participants (not the number of participants without missing values) as the overall participants analyzed.
Time Frame: as for outcome 2
Population: Some participants were not able to complete both conditions of the CSMI test.
Measure: Mean (95% Confidence Interval); unit: unitless (% of sensory system of balance
Arm/Group | Earlier Physical Therapy | Later Physical Therapy (Standard of Care) | Physical Therapy With Home Monitoring | Physical Therapy (Without Home Monitoring)
Number analyzed (Participants) | 82 | 121 | 93 | 110
unitless (% of sensory system of balance
  Estimated Mean Visual Weighting (VS/EO) at Enrollment | 0.134 [0.121 to 0.147] | 0.133 [0.122 to 0.144] | 0.137 [0.124 to 0.150] | 0.130 [0.118 to 0.142]
  Estimated Visual Weighting (VS/EO) Change per Day | -0.0004 [-0.0006 to -0.0002] | -0.0002 [-0.0003 to -0.0001] | -0.00025 [-0.00037 to -0.00013] | -0.00021 [-0.00033 to -0.00009]
  Estimated Mean Vestibular Weighting (SS+VS/EO) at Enrollment | 0.414 [0.393 to 0.435] | 0.415 [0.401 to 0.429] | 0.413 [0.393 to 0.434] | 0.416 [0.400 to 0.432]
  Estimated Vestibular Weighting (SS+VS/EO) Change per Day | 0.0004 [0.0001 to 0.0008] | 0.0004 [0.0002 to 0.0005] | 0.00033 [0.00012 to 0.00054] | 0.00041 [0.00021 to 0.00062]
Statistical Analysis 1: Comparison: Earlier Physical Therapy vs Later Physical Therapy (Standard of Care); Analysis for CSMI Outcome - Visual Weight (VS/EO); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.013, Mixed Models Analysis — a priori threshold p < 0.05; Slope = -0.0003, 95% CI 2-sided [-0.0005 to -0.0001] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Earlier Physical Therapy vs Later Physical Therapy (Standard of Care); Analysis for CSMI Outcome - Vestibular Weight (SS+VS/EO); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.780, Mixed Models Analysis — a priori threshold p < 0.05; Slope = 0.0001, 95% CI 2-sided [-0.0003 to 0.0004] — [estimate comment as in outcome 1, analysis 1]

17. Secondary Outcome: Central Sensorimotor Integration (CSMI) Test: Time Delay
Description: Physical assessment (~45 min) to quantify sway response from a pseudo-random rotating visual surround stimulus on a fixed surface with eyes open (VS/EO) or from combined rotating visual surround and stance surface stimuli (SS+VS/EO) to calculate time delay within the neural controller. We generated inverse probability weights using data from all subjects, thus the overall number of participants (not the number of participants without missing values) as the overall participants analyzed.
Time Frame: as for outcome 2
Population: Some participants were not able to complete both conditions of the CSMI test.
Measure: Mean (95% Confidence Interval); unit: ms
Arm/Group | Earlier Physical Therapy | Later Physical Therapy (Standard of Care) | Physical Therapy With Home Monitoring | Physical Therapy (Without Home Monitoring)
Number analyzed (Participants) | 82 | 121 | 93 | 110
ms
  Estimated Mean Time Delay (VS/EO) at Enrollment | 218.0 [211.5 to 224.5] | 211.0 [206.7 to 215.3] | 213.6 [207.1 to 220.0] | 214.2 [209.2 to 219.2]
  Estimated Time Delay (VS/EO) Change per Day | -0.217 [-0.330 to -0.104] | 0.018 [-0.036 to 0.073] | -0.043 [-0.115 to 0.028] | -0.0257 [-0.095 to 0.043]
  Estimated Mean Time Delay (SS+VS/EO) at Enrollment | 171.0 [165.6 to 176.4] | 170.0 [166.6 to 173.4] | 169.5 [164.6 to 174.4] | 171.9 [167.6 to 176.2]
  Estimated Time Delay (SS+VS/EO) Change per Day | -0.169 [-0.250 to -0.089] | -0.027 [-0.069 to 0.015] | -0.076 [-0.126 to -0.026] | -0.049 [-0.098 to 0.0002]
Statistical Analysis 1: Comparison: Earlier Physical Therapy vs Later Physical Therapy (Standard of Care); Analysis for CSMI Outcome - Time Delay (VS/EO); Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.001, Mixed Models Analysis — a priori threshold p < 0.05; Slope = -0.235, 95% CI 2-sided [-0.361 to -0.110] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Earlier Physical Therapy vs Later Physical Therapy (Standard of Care); Analysis for CSMI Outcome - Time Delay (SS+VS/EO); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.002, Mixed Models Analysis — a priori threshold p < 0.05; Slope = -0.142, 95% CI 2-sided [-0.233 to -0.052] — [estimate comment as in outcome 1, analysis 1]

18. Secondary Outcome: Central Sensorimotor Integration (CSMI) Test: Normalized Stiffness
Description: Physical assessment (~45 min) to quantify sway response from a pseudo-random rotating visual surround stimulus on a fixed surface with eyes open (VS/EO) or from combined rotating visual surround and stance surface stimuli (SS+VS/EO) to calculate normalized stiffness for neural controller. We generated inverse probability weights using data from all subjects, thus the overall number of participants (not the number of participants without missing values) as the overall participants analyzed.
Time Frame: as for outcome 2
Population: Some participants were not able to complete both conditions of the CSMI test.
Measure: Mean (95% Confidence Interval); unit: unitless (%)
Arm/Group | Earlier Physical Therapy | Later Physical Therapy (Standard of Care) | Physical Therapy With Home Monitoring | Physical Therapy (Without Home Monitoring)
Number analyzed (Participants) | 82 | 121 | 93 | 110
unitless (%)
  Estimated Mean Normalized Stiffness (VS/EO) at Enrollment | 1.219 [1.199 to 1.239] | 1.228 [1.211 to 1.245] | 1.212 [1.190 to 1.233] | 1.234 [1.215 to 1.253]
  Estimated Normalized Stiffness (VS/EO) Change per Day | 0.0001 [-0.0004 to 0.0005] | -0.0002 [-0.0004 to -0.000005] | -0.00011 [-0.00036 to 0.00015] | -0.00017 [-0.0042 to 0.00007]
  Estimated Mean Normalized Stiffness (SS+VS/EO) at Enrollment | 1.381 [1.354 to 1.408] | 1.382 [1.362 to 1.402] | 1.373 [1.345 to 1.401] | 1.388 [1.365 to 1.410]
  Estimated Normalized Stiffness (SS+VS/EO) Change per Day | 0.0004 [-0.00002 to 0.0008] | -0.0004 [-0.0005 to -0.0002] | -0.000046 [-0.00030 to 0.00021] | -0.000030 [-0.000055 to -0.000004]
Statistical Analysis 1: Comparison: Earlier Physical Therapy vs Later Physical Therapy (Standard of Care); Analysis for CSMI Outcome - Normalized Stiffness (VS/EO); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.237, Mixed Models Analysis — a priori threshold p < 0.05; Slope = 0.0003, 95% CI 2-sided [-0.0002 to 0.0007] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Earlier Physical Therapy vs Later Physical Therapy (Standard of Care); Analysis for CSMI Outcome - Normalized Stiffness (SS+VS/EO); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.002, Mixed Models Analysis — a priori threshold p < 0.05; Slope = 0.0008, 95% CI 2-sided [0.0003 to 0.001] — [estimate comment as in outcome 1, analysis 1]

19. Secondary Outcome: Central Sensorimotor Integration (CSMI) Test: Normalized Damping
Description: Physical assessment (~45 min) to quantify sway response from a pseudo-random rotating visual surround stimulus on a fixed surface with eyes open (VS/EO) or from combined rotating visual surround and stance surface stimuli (SS+VS/EO) to calculate normalized damping for neural controller. We generated inverse probability weights using data from all subjects, thus the overall number of participants (not the number of participants without missing values) as the overall participants analyzed.
Time Frame: as for outcome 2
Population: Some participants were not able to complete both conditions of the CSMI test.
Measure: Mean (95% Confidence Interval); unit: unitless (%)
Arm/Group | Earlier Physical Therapy | Later Physical Therapy (Standard of Care) | Physical Therapy With Home Monitoring | Physical Therapy (Without Home Monitoring)
Number analyzed (Participants) | 82 | 121 | 93 | 110
unitless (%)
  Estimated Mean Normalized Damping (VS/EO) at Enrollment | 0.469 [0.458 to 0.480] | 0.469 [0.460 to 0.478] | 0.456 [0.445 to 0.466] | 0.479 [0.469 to 0.489]
  Estimated Normalized Damping (VS/EO) Change per Day | 0.0001 [-0.0001 to 0.0003] | -0.0001 [-0.0002 to 0.00005] | 0.000050 [-0.000086 to 0.000186] | -0.00009 [-0.00022 to 0.00004]
  Estimated Mean Normalized Damping (SS+VS/EO) at Enrollment | 0.491 [0.478 to 0.504] | 0.496 [0.485 to 0.507] | 0.485 [0.470 to 0.499] | 0.501 [0.490 to 0.513]
  Estimated Normalized Damping (SS+VS/EO) Change per Day | 0.0002 [-0.00003 to 0.0005] | -0.0002 [-0.0003 to -0.00004] | 0.000015 [-0.000014 to 0.000017] | -0.000011 [-0.000026 to 0.000004]
Statistical Analysis 1: Comparison: Earlier Physical Therapy vs Later Physical Therapy (Standard of Care); Analysis for CSMI Outcome - Normalized Damping (VS/EO); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.247, Mixed Models Analysis — a priori threshold p < 0.05; Slope = 0.0001, 95% CI 2-sided [-0.0001 to 0.0004] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Earlier Physical Therapy vs Later Physical Therapy (Standard of Care); Analysis for CSMI Outcome - Normalized Damping (SS+VSEO); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.008, Mixed Models Analysis — a priori threshold p < 0.05; Slope = 0.0004, 95% CI 2-sided [0.0001 to 0.0007] — [estimate comment as in outcome 1, analysis 1]

20. Secondary Outcome: Central Sensorimotor Integration (CSMI) Test: Evoked CoM Sway
Description: Physical assessment (~45 min) to quantify sway response from a pseudo-random rotating visual surround stimulus on a fixed surface with eyes open (VS/EO) or from combined rotating visual surround and stance surface stimuli (SS+VS/EO) to calculate evoked center-of-mass (CoM) sway. We generated inverse probability weights using data from all subjects, thus the overall number of participants (not the number of participants without missing values) as the overall participants analyzed.
Time Frame: as for outcome 2
Population: Some participants were not able to complete both conditions of the CSMI test.
Measure: Mean (95% Confidence Interval); unit: deg
Arm/Group | Earlier Physical Therapy | Later Physical Therapy (Standard of Care) | Physical Therapy With Home Monitoring | Physical Therapy (Without Home Monitoring)
Number analyzed (Participants) | 82 | 121 | 93 | 110
deg
  Estimated Mean Evoked CoM Sway (VS/EO) at Enrollment | 0.289 [0.256 to 0.322] | 0.281 [0.253 to 0.309] | 0.308 [0.272 to 0.345] | 0.265 [0.236 to 0.294]
  Estimated Evoked CoM Sway (VS/EO) Change per Day | -0.004 [-0.006 to -0.002] | -0.0004 [-0.001 to 0.001] | -0.00029 [-0.00068 to 0.00009] | -0.00014 [-0.00051 to 0.00023]
  Estimated Mean Evoked CoM Sway (SS+VS/EO) at Enrollment | 1.093 [1.027 to 1.159] | 1.068 [1.025 to 1.111] | 1.116 [1.047 to 1.184] | 1.050 [1.003 to 1.096]
  Estimated Evoked CoM Sway (SS+VS/EO) Change per Day | -0.001 [-0.002 to -0.0003] | 0.0002 [-0.0002 to 0.001] | -0.00036 [-0.00098 to 0.00026] | -0.00049 [-0.00066 to 0.00056]
Statistical Analysis 1: Comparison: Earlier Physical Therapy vs Later Physical Therapy (Standard of Care); Analysis for CSMI Outcome - Evoked Center of Mass (CoM) Sway (VS/EO); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.003, Mixed Models Analysis — a priori threshold p < 0.05; Slope = -0.004, 95% CI 2-sided [-0.006 to -0.001] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Earlier Physical Therapy vs Later Physical Therapy (Standard of Care); Analysis for CSMI Outcome - Evoked CoM Sway (SS+VS/EO); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.004, Mixed Models Analysis — a priori threshold p < 0.05; Slope = -0.001, 95% CI 2-sided [-0.003 to -0.0005] — [estimate comment as in outcome 1, analysis 1]

21. Secondary Outcome: Central Sensorimotor Integration (CSMI) Test: Internal Sensory Noise
Description: Physical assessment (~45 min) to quantify sway response from a pseudo-random rotating visual surround stimulus on a fixed surface with eyes open (VS/EO) or from combined rotating visual surround and stance surface stimuli (SS+VS/EO) to internal sensory noise. We generated inverse probability weights using data from all subjects, thus the overall number of participants (not the number of participants without missing values) as the overall participants analyzed.
Time Frame: as for outcome 2
Population: Some participants were not able to complete both conditions of the CSMI test.
Measure: Mean (95% Confidence Interval); unit: deg
Arm/Group | Earlier Physical Therapy | Later Physical Therapy (Standard of Care) | Physical Therapy With Home Monitoring | Physical Therapy (Without Home Monitoring)
Number analyzed (Participants) | 82 | 121 | 93 | 110
deg
  Estimated Mean Internal Sensory Noise (VS/EO) at Enrollment | 0.088 [0.079 to 0.097] | 0.087 [0.079 to 0.095] | 0.092 [0.081 to 0.104] | 0.084 [0.076 to 0.091]
  Estimated Internal Sensory Noise (VS/EO) Change per Day | -0.003 [-0.006 to -0.0004] | 0.0002 [-0.001 to 0.002] | 0.000054 [-0.00011 to 0.00022] | -0.000051 [-0.00021 to 0.00010]
  Estimated Mean Internal Sensory Noise (SS+VS/EO) at Enrollment | 0.136 [0.125 to 0.147] | 0.126 [0.117 to 0.135] | 0.135 [0.123 to 0.147] | 0.127 [0.116 to 0.137]
  Estimated Internal Sensory Noise (SS+VS/EO) Change per Day | -0.003 [-0.005 to -0.001] | -0.0005 [-0.001 to 0.001] | 0.0000097 [-0.0000172 to 0.0000192] | -0.00030 [-0.00037 to -0.00027]
Statistical Analysis 1: Comparison: Earlier Physical Therapy vs Later Physical Therapy (Standard of Care); Analysis for CSMI Outcome - Internal Sensory Noise (VS/EO); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.031, Mixed Models Analysis — a priori threshold p < 0.05; Slope = -0.004, 95% CI 2-sided [-0.007 to -0.0003] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Earlier Physical Therapy vs Later Physical Therapy (Standard of Care); Analysis for CSMI Outcome - Internal Sensory Noise (SS+VS/EO); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.003, Mixed Models Analysis — a priori threshold p < 0.05; Slope = -0.003, 95% CI 2-sided [-0.005 to -0.0003] — [estimate comment as in outcome 1, analysis 1]

22. Other Pre Specified Outcome: Post-concussion Symptom Scale From the Sport Concussion Assessment (SCAT) Tool Version 5
Description: A weekly questionnaire assessing mTBI symptom severity over 14 weeks with 22 items rated from 0 (none) to 6 (severe). Total symptom severity score out of 132. High scores indicate worse performance.
Time Frame: Collected weekly throughout study duration (week 0 to week 14).
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Earlier Physical Therapy | Later Physical Therapy (Standard of Care) | Physical Therapy With Home Monitoring | Physical Therapy (Without Home Monitoring)
Number analyzed (Participants) | 82 | 121 | 93 | 110
score on a scale
  Estimated Mean at Enrollment | 56.5 [51.9 to 61.2] | 58.8 [54.7 to 62.8] | 59.0 [54.4 to 63.5] | 56.9 [52.8 to 61.1]
  Estimated Change per Day | -0.349 [-0.398 to -0.300] | -0.317 [-0.358 to -0.276] | -0.361 [-0.414 to -0.308] | -0.313 [-0.374 to -0.252]
Statistical Analysis 1: Comparison: Earlier Physical Therapy vs Later Physical Therapy (Standard of Care); Test type: Other — Linear mixed effect model containing fixed effects for group (earlier or later), time since injury, and group x time since injury interaction with random intercepts, covariates (age and gender), and inverse probability weights. Later Physical Therapy Group served as the reference; p = 0.3221, Mixed Models Analysis — a priori threshold p < 0.05; Slope = -0.0321, 95% CI 2-sided [-0.0957 to 0.0315] — [estimate comment as in outcome 1, analysis 1]

23. Other Pre Specified Outcome: Insomnia Severity Index (ISI)
Description: Self-rated questionnaire (~5 minutes) to rate sleep as a potential covariate for recovery rated on a 5-point scale (0: none; 4: very severe) with a maximum score of 28. High scores indicate worse outcomes.
Time Frame: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Earlier Physical Therapy | Later Physical Therapy (Standard of Care) | Physical Therapy With Home Monitoring | Physical Therapy (Without Home Monitoring)
Number analyzed (Participants) | 82 | 121 | 93 | 110
score on a scale
  Estimated Mean at Enrollment | 14.0 [12.7 to 15.3] | 16.1 [15.0 to 17.2] | 15.5 [14.2 to 16.8] | 15.0 [13.9 to 16.2]
  Estimated Change per Day | -0.0725 [-0.0977 to -0.0473] | -0.0590 [-0.0705 to -0.0474] | -0.060 [-0.076 to -0.045] | -0.059 [-0.073 to -0.044]
Statistical Analysis 1: Comparison: Earlier Physical Therapy vs Later Physical Therapy (Standard of Care); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.336, Mixed Models Analysis — a priori threshold p < 0.05; Slope = -0.0136, 95% CI 2-sided [-0.0413 to 0.0142] — [estimate comment as in outcome 1, analysis 1]

24. Other Pre Specified Outcome: Head Impact Test (HIT) - 6
Description: Self-rated questionnaire (~5 minutes of 6 items to rate headache severity as a potential covariate for recovery rated on a 5-point scale (6: never; 13: always) with a maximum score of 78. High scores indicate worse outcomes.
Time Frame: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Earlier Physical Therapy | Later Physical Therapy (Standard of Care) | Physical Therapy With Home Monitoring | Physical Therapy (Without Home Monitoring)
Number analyzed (Participants) | 82 | 121 | 93 | 110
score on a scale
  Estimated Mean at Enrollment | 61.7 [60.3 to 63.2] | 62.5 [61.4 to 63.7] | 62.4 [61.0 to 63.8] | 62.0 [60.8 to 63.2]
  Estimated Change per Day | -0.123 [-0.156 to -0.0885] | -0.0819 [-0.0975 to -0.0663] | -0.110 [-0.130 to -0.090] | -0.076 [-0.096 to -0.056]
Statistical Analysis 1: Comparison: Earlier Physical Therapy vs Later Physical Therapy (Standard of Care); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.033, Mixed Models Analysis — a priori threshold p < 0.05; Slope = -0.0406, 95% CI 2-sided [-0.0779 to -0.0032] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Study duration (week 0 to week 14)
Arm/Group | Earlier Physical Therapy | Later Physical Therapy (Standard of Care) | Physical Therapy With Home Monitoring | Physical Therapy (Without Home Monitoring)
All-Cause Mortality (participants affected / at risk) | 0/82 | 0/121 | 0/93 | 0/110
Serious Adverse Events (participants affected / at risk) | 0/82 | 0/121 | 0/93 | 0/110
Other Adverse Events (participants affected / at risk) | 3/82 | 0/121 | 2/93 | 1/110
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Earlier Physical Therapy (N=82) | Later Physical Therapy (Standard of Care) (N=121) | Physical Therapy With Home Monitoring (N=93) | Physical Therapy (Without Home Monitoring) (N=110)
Medical Event: Nose bleed (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) — Subject reported getting a blood nose after completing their home exercise program. This was a one time occurrence, mild intensity, causality was unrelated and resolved the day it occurred. The subject remained in the study
Medical Event: Swelling of Eye (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — Reported eye swelling following home exercise program. Resolved the same day is occurred, mild intensity, cause was unrelated to study, no medical attention required and remained in study.
Discomfort While Testing (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — Participant leg hit the side/arm of the chair during rotary chair testing. This resolved the same day it occurred, was mild intensity, related to the study and the subject remained in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-07-08): https://cdn.clinicaltrials.gov/large-docs/41/NCT03479541/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-17): https://cdn.clinicaltrials.gov/large-docs/41/NCT03479541/SAP_001.pdf